CLINICAL TRIAL: NCT02817906
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of ITI-007 in the Treatment of Agitation in Patients With Dementia, Including Alzheimer's Disease
Brief Title: ITI-007 for the Treatment of Agitation in Patients With Dementia, Including Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pre-specified Interim Analysis Indicated Futility
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-201
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Agitation in Dementia, Including Alzheimer's Disease
MeSH Terms: conditions — Aberrant Motor Behavior in Dementia | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ITI-007 (Experimental): 9 mg ITI-007 administered as a solid oral dose formulation once daily for 4 weeks.
  Interventions: Drug: ITI-007
- Placebo (Placebo Comparator): Placebo administered as a visually-matched solid oral dose formulation once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-007
  Arms: ITI-007
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study comparing the efficacy and safety of ITI-007 versus placebo administered orally once daily in the treatment of agitation in patients with dementia, including Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Alzheimer's disease
* Clinically significant symptoms of agitation secondary to probable Alzheimer's disease
* Able to attend outpatient clinic visits with primary caregiver

Exclusion Criteria:

* Unable to comply with study procedures
* Considered medically inappropriate for study participation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kozauer, M.D., Study Director — Intra-Cellular Therapies, Inc.
Locations (26):
- United States (26):
  - Sun City, Arizona
  - Little Rock, Arkansas
  - Rogers, Arkansas
  - Costa Mesa, California
  - Glendale, California
  - Irvine, California
  - Lemon Grove, California
  - Long Beach, California
  - Oceanside, California
  - Riverside, California
  - Santa Ana, California
  - Hallandale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Orlando, Florida
  - Suwanee, Georgia
  - Honolulu, Hawaii
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Marlton, New Jersey
  - Toms River, New Jersey
  - Brooklyn, New York
  - Staten Island, New York
  - Centerville, Ohio
  - Dayton, Ohio
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ITI-007 9 mg: 9 mg ITI-007 administered as a solid oral dose formulation once daily for 4 weeks.
  ITI-007(lumateperone tosylate) 9 mg is equivalent to 6 mg lumateperone, the free base or active moiety.
Period: Overall Study
Arm/Group | ITI-007 9 mg | Placebo
Started (Part A-Number of subjects treated) | 86 (87 patients were randomized but only 86 received study drug. The number completed and discontinued is based on the 86 patients that received study drug.) | 89 (90 patients were randomized but only 89 received study drug. The number completed and discontinued is based on 89 patients that received study drug.)
Completed (Part A) | 70 | 84
Not Completed | 16 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Study Terminated by Sponsor | 2 | 2
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- 9 mg ITI-007: 9 mg ITI-007 administered as a solid oral dose formulation once daily for 4 weeks
- Total: Total of all reporting groups
Arm/Group | 9 mg ITI-007 | Placebo | Total
Number analyzed (Participants) | 86 | 89 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (8.64) | 74.1 (8.61) | 74.8 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 57 | 101
  Male | 42 | 32 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 75 | 148
  Black or African American | 10 | 10 | 20
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Multiple | 0 | 1 | 1
  Unknown | 0 | 1 | 1
CMAI-C [Mean (Standard Deviation); unit: units on a scale] — The Cohen-Mansfield Agitation Inventory-Community Version is a 37-item scale for identifying and quantifying agitated behaviors in elderly persons in a community setting. Each item is rated from 1='Never' to 7='Several Times Per Hour'. Each category contains a pre-specified subset of the CMAI-C items. The score of each category is the sum of the CMAI-C items included in that category: Aggressive Behavior-Sum of 9 CMAI-C items, ranges from 9 to 63; Non-Aggressive Agitated Behavior-Sum of 6 CMAI-C items, ranges from 6 to 42; Verbally Agitated Behavior-Sum of 4 CMAI-C items, ranges from 4 to 28.
  units on a scale
    CMAI-C Aggressive Behavior | 13.28 (4.51) | 14.08 (5.92) | 13.69 (5.27)
    CMAI-C Non-Aggressive Agitated Behavior | 17.20 (7.42) | 17.46 (7.05) | 17.33 (7.22)
    CMAI-C Verbally Agitated Behavior | 15.37 (4.95) | 15.65 (5.02) | 15.51 (4.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Cohen-Mansfield Agitation Inventory - Community Version (CMAI-C)
Description: The Cohen-Mansfield Agitation Inventory-Community Version is a 37-item scale for identifying and quantifying agitated behaviors in elderly persons in a community setting. Each item is rated from 1='Never' to 7='Several Times Per Hour'. Each category contains a pre-specified subset of the CMAI-C items. The score of each category is the sum of the CMAI-C items included in that category: Aggressive Behavior-Sum of 9 CMAI-C items, ranges from 9 to 63; Non-Aggressive Agitated Behavior-Sum of 6 CMAI-C items, ranges from 6 to 42; Verbally Agitated Behavior-Sum of 4 CMAI-C items, ranges from 4 to 28.
Time Frame: 4 weeks (28 Days)
Population: Intent-to-Treat Set (Study stopped for futility)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 9 mg ITI-007 | Placebo
Number analyzed (Participants) | 78 | 84
score on a scale
  Aggressive Agitated Behavior | -1.0 (0.37) | -2.3 (0.33)
  Non-Aggressive Agitated Behavior | -4.1 (0.72) | -3.9 (0.65)
  Verbally Agitated Behavior | -2.9 (0.49) | -2.3 (0.45)

2. Secondary Outcome: Change From Baseline in the Clinical Global Impression Scale for Severity of Illness (CGI-S)
Description: The CGI scale for Severity of Illness is a standardized assessment tool to rate the overall severity of illness and efficacy of medication. CGI-S of Agitation and CGI-S of Aggression will be used in this study as a measure of efficacy.
  Scores on the CGI-S range from 1 (not ill at all) to 7 (among the most extremely ill).
Time Frame: 4 weeks (28 Days)
Population: Intent-to Treat Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 9 mg ITI-007 | Placebo
Number analyzed (Participants) | 78 | 84
score on a scale
  CGI-S Aggression | -0.4 (0.12) | -0.6 (0.10)
  CGI-S Agitation | -0.8 (0.11) | -0.9 (0.10)

ADVERSE EVENTS:
Time Frame: 4 weeks of double blind treatment.
Description: Safety Analysis Set
Arm/Group | 9 mg ITI-007 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/89
Serious Adverse Events (participants affected / at risk) | 2/86 | 1/89
Other Adverse Events (participants affected / at risk) | 13/86 | 8/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9 mg ITI-007 (N=86) | Placebo (N=89)
Urinary tract infection (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Ammonia Increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 9 mg ITI-007 (N=86) | Placebo (N=89)
Dizziness (Nervous system disorders) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Somnolence (Nervous system disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
CMAI-C Factor Composite score (Aggressive Behavior, Non-Aggressive Agitated Behavior, Verbally Agitated Behavior) was the primary efficacy measure not the CMAI-C Total score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT02817906/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT02817906/SAP_001.pdf